CLINICAL TRIAL: NCT02431897
Title: Investigation to Minimize Prolapse Recurrence of the Vagina Using Estrogen
Acronym: IMPROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other); Women and Infants Hospital of Rhode Island (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, David Rahn, MD, Associate Professor, Dept. of Obstetrics & Gynecology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 022015-117
Record Dates: First submitted 2015-04-23; First posted 2015-05-01 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Pelvic Organ Prolapse; Urogenital Prolapse; Vaginal Vault Prolapse; Cystocele; Uterine Prolapse; Vaginal Prolapse; Pelvic Floor Disorders
Keywords: Pelvic Organ Prolapse; Pelvic Floor Disorders; Therapy, Estrogen Replacement; Estrogens, Conjugated
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Uterine Prolapse; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estrogen Cream (Experimental): Conjugated Estrogens cream
  Interventions: Drug: Conjugated Estrogens Cream
- Placebo Cream (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Conjugated Estrogens Cream — 0.625mg/1g cream, 1g applied vaginally nightly for 2 weeks then 2x/week for >5 weeks before surgery, then 2x/week for 1 year after surgery.
  Other Names: Premarin Vaginal Cream
  Arms: Estrogen Cream
Drug: Placebo Cream — 1g applied vaginally nightly for 2 weeks then 2x/week for >5 weeks before surgery, then 2x/week for 1 year after surgery.
  Arms: Placebo Cream

SUMMARY:
This study randomizes postmenopausal women with symptomatic pelvic organ prolapse planning native tissue transvaginal surgical repair to 6-8 weeks of preoperative and 1-year continued postoperative vaginal estrogen cream compared to placebo cream. This clinical trial and basic science investigation are designed to understand the mechanisms by which local estrogen treatment affects connective tissues of the pelvic floor and determine whether its use before and after prolapse repair will (i) improve success rates of the surgical intervention and minimize prolapse recurrence and (ii) impact favorably upon symptoms of other pelvic floor disorders.

DETAILED DESCRIPTION:
This is a double-blind randomized trial of intravaginal estrogen (conjugated estrogens, 0.625mg/1g cream) vs. placebo in postmenopausal women (up to n=222 enrolled and randomized in order for 188 to undergo surgery) with symptomatic prolapse beyond the hymen planning transvaginal native tissue repairs. Medication will be started >5 weeks before surgery and continued for 1 year postoperatively, i.e. until scar remodeling is complete. The investigators aim to determine if pre- and postoperative intravaginal estrogen therapy (i) results in anatomic and patient-reported subjective improvement in pelvic organ support, and (ii) impacts other pelvic floor disorders (overactive bladder and incontinence, sexual function and pain, postoperative cystitis), satisfaction, quality of life, and vaginal wound healing. Finally, (iii) the investigators will determine the potential mechanisms by which local estrogen treatment alters pelvic organ support by examining full-thickness vaginal wall biopsies taken at the time of surgery for histologic, connective tissue, and smooth muscle synthesis and degradative changes. The investigators expect this will highlight other novel targets for future therapies in prolapse repair and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal: no menses for >1 year
* Minimum age: 48 years
* Symptomatic apical and/or anterior vaginal wall prolapse, stage 2 or greater
* No estrogen replacement within the last month (may come off current treatment, i.e. wash out, to join the study)
* Medically fit for elective surgery
* Physically able to apply/insert the study drug
* Available for clinic follow-up for minimum 1yr

Exclusion Criteria:

* Concurrent use of steroid creams for other indications (e.g. lichen sclerosis)
* BMI >35 kg/m2
* Recent history (within last month) of vaginal infection or vaginitis
* Contraindications to estrogen therapy (e.g. spontaneous DVT, stroke, breast or endometrial/ hormone-responsive cancer, genital bleeding of unknown cause)
* History of connective tissue disease
* Any oral or transdermal estrogen, SERM, or other medication impacting vaginal milieu
* History of vaginal irradiation
* Allergy to Premarin or its constituents
* Prior apical repair or use of mesh for prolapse repair
* Current tobacco use

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D Rahn, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Rahn DD, Richter HE, Sung VW, Larsen WI, Hynan LS. Design of a Randomized Clinical Trial of Perioperative Vaginal Estrogen Versus Placebo With Transvaginal Native Tissue Apical Prolapse Repair (Investigation to Minimize Prolapse Recurrence of the Vagina using Estrogen: IMPROVE). Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):e227-e233. doi: 10.1097/SPV.0000000000000899. PMID 32541299
- [Derived] Rahn DD, Richter HE, Sung VW, Pruszynski JE. Three-year outcomes of a randomized clinical trial of perioperative vaginal estrogen as adjunct to native tissue vaginal apical prolapse repair. Am J Obstet Gynecol. 2024 Aug;231(2):263.e1-263.e10. doi: 10.1016/j.ajog.2024.04.042. Epub 2024 May 4. PMID 38710269
- [Derived] Rahn DD, Richter HE, Sung VW, Hynan LS, Pruszynski JE. Characteristics Associated With Surgical Failure After Native Tissue Apical Prolapse Repair. Obstet Gynecol. 2024 Feb 1;143(2):312-319. doi: 10.1097/AOG.0000000000005478. Epub 2023 Dec 7. PMID 38061041
- [Derived] Rahn DD, Richter HE, Sung VW, Pruszynski JE, Hynan LS. Perioperative Vaginal Estrogen as Adjunct to Native Tissue Vaginal Apical Prolapse Repair: A Randomized Clinical Trial. JAMA. 2023 Aug 15;330(7):615-625. doi: 10.1001/jama.2023.12317. PMID 37581673
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855
- [Derived] Rahn DD, Richter HE, Sung VW, Hynan LS, Pruszynski JE. Effects of preoperative intravaginal estrogen on pelvic floor disorder symptoms in postmenopausal women with pelvic organ prolapse. Am J Obstet Gynecol. 2023 Sep;229(3):309.e1-309.e10. doi: 10.1016/j.ajog.2023.05.023. Epub 2023 May 25. PMID 37244454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 206 participants consented/enrolled, 7 were not randomized: 4 withdrew consent before randomization, and 3 were found to be ineligible and were not randomized. This left n=199 for randomization.
Period: Overall Study
Arm/Group | Estrogen Cream | Placebo Cream
Started | 102 | 97
Completed | 93 | 93
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estrogen Cream | Placebo Cream | Total
Number analyzed (Participants) | 102 | 97 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (6.1) | 65.2 (7.3) | 65.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 97 | 199
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 78 | 73 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 92 | 89 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Gravidity [Median (Inter-Quartile Range); unit: pregnancies] | 3 [2 to 3] | 2 [2 to 3] | 3 [2 to 3]
Vaginal deliveries [Median (Inter-Quartile Range); unit: births] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Surgical "Failure" Defined by (i) Anatomic Assessment of Prolapse, (ii) Presence of Bulge Symptoms, and/or (Iii) Retreatment of Prolapse
Description: Cumulative failures, as measured by (i) anatomic assessment of prolapse, (ii) presence of bulge symptoms, and/or (iii) retreatment of pelvic organ prolapse
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
Participants | 18 | 8

2. Secondary Outcome: Condition Specific (i.e. Pelvic Organ Prolapse) Symptom Bother as Measured by Pelvic Floor Distress Inventory-20 (PFDI-20) Questionnaire
Description: Questionnaire score at 12 months in overall condition-specific symptom bother as measured by Pelvic Floor Distress Inventory-20 (PFDI-20) questionnaire, which is scored from 0-300, higher scores being worse (i.e., more distressing)
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 23.1 (4.6) | 23.1 (4.7)

3. Secondary Outcome: Condition Specific (i.e. Pelvic Organ Prolapse) Quality of Life as Measured by Pelvic Floor Impact Questionnaire-7 (PFIQ-7)
Description: Questionnaire score at 12 months in overall condition-specific quality of life as measured by Pelvic Floor Impact Questionnaire-7 (PFIQ-7) questionnaire, which is scored from 0-300, higher scores being worse (i.e., more distressing)
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 8.9 (4.5) | 9.5 (4.6)

4. Secondary Outcome: Generic Quality of Life as Measured by SF-12 Questionnaire
Description: Generic (physical component) quality of life as measured by SF-12 questionnaire at 12 months. Scores range from 0-100, with higher scores indicating better physical functioning; the US population average is 50 points.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 52.1 (0.9) | 53.2 (0.9)

5. Secondary Outcome: Urinary Symptoms as Measured by Urinary Subscale Questions of the Pelvic Floor Distress Inventory-20 (PFDI-20) Questionnaire, i.e. the Urinary Distress Inventory, UDI-6
Description: Urinary symptom bother as measured by urinary subscale questions of the Pelvic Floor Distress Inventory-20 (PFDI-20) questionnaire, i.e. the Urinary Distress Inventory, UDI-6. This is scored from 0-100, with greater scores indicating greater symptom bother.
Time Frame: Time of surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 102 | 97
score on a scale | 38.2 (2.7) | 37.7 (2.8)

6. Secondary Outcome: Urinary Symptoms as Measured by Urinary Subscale Questions of the Pelvic Floor Distress Inventory-20 (PFDI-20) Questionnaire, i.e. the Urinary Distress Inventory, UDI-6
Description: as for outcome 5
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 9.8 (2.1) | 9.2 (2.2)

7. Secondary Outcome: Urinary Symptoms as Measured by Urinary Subscale Questions of the Pelvic Floor Impact Questionnaire (PFIQ-7), i.e. the Urinary Impact Questionnaire
Description: Urinary symptom impact on quality of life as measured by urinary subscale questions of the Pelvic Floor Impact Questionnaire (PFIQ-7), i.e. the Urinary Impact Questionnaire. This is scored from 0-100, with greater scores indicating worse impact on quality of life.
Time Frame: Time of surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 102 | 97
score on a scale | 26.9 (1.8) | 25.2 (1.8)

8. Secondary Outcome: Urinary Symptoms as Measured by Urinary Subscale Questions of the Pelvic Floor Impact Questionnaire (PFIQ-7), i.e. the Urinary Impact Questionnaire
Description: as for outcome 7
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 1.2 (1.9) | 2.6 (1.9)

9. Secondary Outcome: Sexual Function as Measured by the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR)
Description: Sexual function in sexually-active women as measured by the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). The score ranges from 1 (worse sexual experience) to 5 (better sexual experience) with midrange scores commonly seen in women with pelvic floor disorders.
Time Frame: Time of surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 102 | 97
score on a scale | 3.13 (0.10) | 3.12 (0.10)

10. Secondary Outcome: Sexual Function as Measured by the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR)
Description: as for outcome 9
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 93 | 93
score on a scale | 3.55 (0.10) | 3.70 (0.10)

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants reporting any adverse events from baseline randomization to 12 months postoperatively
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Estrogen Cream | Placebo Cream
Number analyzed (Participants) | 102 | 97
Participants | 73 | 68

ADVERSE EVENTS:
Time Frame: From baseline randomization to 12 months postoperatively
Arm/Group | Estrogen Cream | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/97
Serious Adverse Events (participants affected / at risk) | 10/102 | 11/97
Other Adverse Events (participants affected / at risk) | 56/102 | 51/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Cream (N=102) | Placebo Cream (N=97)
Trimalleolar fracture, closed (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Anaphylactic shock due to adverse food reaction (Immune system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Fractured hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection MRSA (Infections and infestations) | 1 (1) | 0 (0)
Carcinoma breast stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3)
Viral infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bladder injury (Surgical and medical procedures) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac catheter ablation (Cardiac disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Cream (N=102) | Placebo Cream (N=97)
Urinary tract infection (Infections and infestations) | 18 (20) | 22 (32)
Yeast infection (Infections and infestations) | 10 (10) | 6 (6)
Nausea and vomiting (Gastrointestinal disorders) | 7 (7) | 6 (6)
Dyspareunia (Reproductive system and breast disorders) | 6 (6) | 5 (5)
Granulation tissue (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Vaginal itching (Reproductive system and breast disorders) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02431897/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02431897/ICF_001.pdf